CLINICAL TRIAL: NCT02499250
Title: Effect of Daily Remote Ischemic Conditioning on the Life Quality of Refractory Angina Pectoris Patients and the Mechanism
Brief Title: Effect of Daily Remote Ischemic Conditioning on the Life Quality of Refractory Angina Pectoris Patients
Acronym: D-RIC-RAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Li Zhao MD,PhD, attending physician, Navy General Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HZKY-PJ-2014-1-A
Record Dates: First submitted 2015-06-21; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Refractory Angina Pectoris
Keywords: refractory angina pectoris; remote ischemic conditioning; life quality; anxiety; depression; inflammation
MeSH Terms: conditions — Angina Pectoris; Anxiety Disorders; Depression; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC arm (Experimental): The subjects will be interviewed and have their baseline frequency and severity of angina pectoris recorded, then they will receive daily remote ischemic conditioning plus optimal medical treatment over 30 days.
  Interventions: Device: remote ischemic conditioning (TDFT-12-A2); Drug: Optimal medical treatment
- Control arm (Active Comparator): The subjects will be interviewed and have their baseline frequency and severity of angina pectoris recorded, then they will receive optimal medical treatment over 30 days.
  Interventions: Drug: Optimal medical treatment

INTERVENTIONS:
Device: remote ischemic conditioning (TDFT-12-A2) — The subjects will receive twice daily of 4×5min/5min ischemic/reperfusion of both arms (remote ischemic conditioning) over 30 days using the "TDFT-12-A2" device produced by "Shenzhen TDF Tai Smart technology Co., Ltd."
  Other Names: RIC
  Arms: RIPC arm
Drug: Optimal medical treatment — The subjects will receive optimal medical treatment according up-to-date guidelines, including adequate antiplatelet therapy, statins, β-blocker and nitrates, plus angiotensin converting enzyme inhibitor(ACEI)/angiotensin receptor blocker(ARB),oral anticoagulants, if necessary.
  Other Names: OMT

SUMMARY:
The purpose is to test whether daily ischemic conditioning of the arms over 30 days could reduce the frequency and severity of angina pectoris and improve the life quality of refractory angina pectoris patients.

DETAILED DESCRIPTION:
Refractory angina pectoris denotes "chronic stable angina that persists despite optimal medication and when revascularisation is unfeasible or where the risks are unjustified". These patients could potentially be relieved by non-conventional treatments like remote ischemic conditioning, and actually this effect has been observed in several cases in the center of the sponsor. This study is a pilot study to measure the efficacy and safety of this method in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed angina pectoris that remains despite optimal medical treatment;
* No chance of further revascularization or refusal to do revascularization;
* The frequency and Canadian Cardiovascular Society (CCS) scale stays stable over the past 3 months before inclusion.

Exclusion Criteria:

* Known or highly suspected abnormality of peripheral arteries, veins, or extremities;
* Infection or fever in the past month;
* Blood pressure over 180/110 millimeters of mercury (mmHg) or below 80/50mmHg;
* Refusal to comply with the study protocol;
* Currently under sulfonylureas or prostaglandins therapy;
* Other conditions that the researchers judge as inappropriate to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Frequencies of angina pectoris onset | 30 days
  The total times of angina pectoris onset over one week
Canadian Cardiovascular Society Angina Class | 30 days
  Ranging from class 1 to class 4 according to its definition

SECONDARY OUTCOMES:
Flow mediated vasodilation in percentage increase | 30 days
  Reported as percent increase of brachial artery diameter induced by release of the forearm after ligation, accessed by experienced ultrasound professional.
Flow mediated vasodilation in absolute increase | 30 days
  Reported as absolute increase (cm) of brachial artery diameter induced by release of the forearm after ligation, accessed by experienced ultrasound professional.
Self-Rating Anxiety Scale | 30 days
  Reported as the Self-Rating Anxiety score
Self-Rating Depression Scale | 30 days
  Reported as the Self-Rating Depression score
Inflammatory cytokines expression | 30 days
  Reported as the serum levels of inflammatory cytokines measured by ELISA kits, including tumor necrosis factor(TNF-α)，Interleukine(IL)-6，and IL-10; The expression of signaling proteins in separated blood mononuclear cells,including hypoxia inducible factor(HIF) 1α.
Grip strength | 30 days
  Measured by a simple Grip strength meter (CAMRY) and reported as kilograms of strength.
Skin and muscle abnormalities | 1,7 and 30 days
  Whether or not the skin of the arm has bruises, and whether or not the arm has sore or pain feeling.
Circulating CD34+ progenitor cells | 30 days
  The percent of circulating cluster of differentiation(CD)34+ progenitor cells in separated mononuclear cells measured by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Tianchang Li, MD, PhD, Study Chair — Heart center, Navy General Hospital
Locations (1):
- Heart Center, Navy General Hospital of PLA, Beijing, Beijing Municipality, China